CLINICAL TRIAL: NCT05549284
Title: a Single Arm,Multi-center,Phase II Clinical Trial of Combined Therapy for Orelabrutinib,Rituximab and Methotrexate(RMO)in Newly-diagnosed Primary Center Nervous System Lymphoma(PCNSL)
Brief Title: Orelabrutinib,Rituximab and Methotrexate in Newly-diagnosed Primary Central Nervous System Lymphoma(PCNSL)
Acronym: RMO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-947168-88
Record Dates: First submitted 2022-08-24; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Primary Central Nervous System Lymphoma
MeSH Terms: interventions — orelabrutinib; Rituximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orelabrutinib,Rituximab and Methotrexate (Experimental): Rituximab 375 mg/m2 d1; MTX 3.5mg/m2,d2; Orelabrutinib 150g/day; every three week/cycle.
  Interventions: Drug: Orelabrutinib,Rituximab and Methotrexate

INTERVENTIONS:
Drug: Orelabrutinib,Rituximab and Methotrexate — Orelabrutinib, Rituximab combined with high-dose Methotrexate(RMO) as first line regimens in the treatments of newly diagnosed primary central nervous system lymphoma. The response will be evaluated every 2 cycles. Patients who achieved complete remission (CR) or partial remission (PR) will receive further treatment, and there are 6 cycles of RMO regimen for the induction. The patients with stable disease (SD) or progressed disease(PD) will withdraw from the trial and receive salvage regimens. After total 6 induction cycles, the investigators evaluate the efficiency again. After 6 cycles, the patients who receive CR or PR, can tolerate Autologous Hematopoietic Stem Cell Transplantation (AHSCT) will be candidates of high-dose chemotherapy and stem rescue. The patients who achieve CR or PR, cannot tolerate AHSCT will go to whole brain radiotherapy or Orelabrutinib maintenance. The patients with SD or PD will receive salvage regimen.
  Other Names: RMO

SUMMARY:
This is a prospective single arm,multi-center,phase 2 study,and this study is to evaluate the efficacy and safety of Orelabrutinib,Rituximab combined with high-dose Methotrexate(RMO) as first line regimens in the treatments of newly diagnosed primary central nervous system lymphoma(PCNSL).Objective response and complete response are the primary endpoint.

DETAILED DESCRIPTION:
This is a single-arm,multicenter,phase 2 study to evaluate the efficacy and safety of Orelabrutinib,Rituximab combined with high-dose Methotrexate(RMO) as first line regimens in the treatments of newly diagnosed primary central nervous system lymphoma.The response will be evaluated every 2 cycles.Patients who achieved complete remission(CR) or partial remission(PR) will receive further treatment,and there are 6 cycles of RMO regimen for the induction.The patients with stable disease(SD) or progressed disease(PD) will withdraw from the trial and receive salvage regimens.After total 6 induction cycles,the investigators evaluate the efficiency again.After 6 cycles,the patients who receive CR or PR,can tolerate Autologous Hematopoietic Stem Cell Transplantation(AHSCT) will be candidates of high-dose chemotherapy and stem rescue.The patients who achieve CR or PR,cannot tolerate AHSCT will go to whole brain radiotherapy or Orelabrutinib maintenance.The patients with SD or PD will receive salvage regimen.

ELIGIBILITY:
Inclusion Criteria:

* primary central nervous system diffuse large B-cell lymphoma histologically confirmed by brain biopsy;
* Aged 18-70 years
* Signature of informed consent;
* At least one measurable lesion;
* Neutropile≥1.5X109/L,Hemoglobin≥80g/L,Platelets≥75X109/L,Billrubin<2XULN,ALT<4XULN,AST4XULN
* The expected survival time is at least 3 months

Exclusion Criteria:

* Those who have contraindications to any of the components in the Orelabrutinib,Rituximab and HD-MTX
* History of other malignancies that may affect the compliance of the research protocol or the analysis of the results
* Severe cardiac insufficiency
* Other antitumor treatments were used
* Human immunodeficiency virus(HIV)antibody is positive
* Pregnant or lactating women
* Researchers consider if anyone not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
primary endpoint | Enrollment is expected to last for two year, followed up for five years
  Objective response rate(ORR) is the primary endpoint

SECONDARY OUTCOMES:
secondary endpoints | Enrollment is expected to last for two year, followed up for five years
  Complete rate(CR)、progression free survival(PFS)、overall survival(OS) are the secondary endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital 307, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No